## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

## Study information

| Title | Assessment of 13-valent pneumococcal conjugate |
|---|---|
| | vaccine effectiveness among people with HIV in the<br>United States |
| Protocol number | B1851217 |
| Protocol version identifier | 3.0 |
| Date | 06 December 2023 |
| Active substance | |
| Medicinal product | Prevnar 13 |
| Research question and objectives | <ol> <li>The primary objectives include: <ol> <li>Estimate vaccine effectiveness (VE) of PCV13 for invasive pneumococcal disease (IPD) among people living with HIV (PLWH) ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up</li> </ol> </li> <li>Estimate VE of PCV13 for pneumococcal pneumonia among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up</li> <li>Estimate VE of PCV13 for all-cause pneumonia among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of overall and, if feasible, at 3, 5, and 7 years of</li> </ol> |
| | follow-up The secondary objectives of this study are to estimate: 1. Estimate VE of PCV13 for pneumococcal pneumonia or pneumonia with unspecified causes among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up 2. Estimate VE of PCV13 for pneumonia with unspecified causes among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up |

| Author | PPD | , PhD, MPH |
|--------|--------------|------------|
| | Pfizer, Inc. | _ |
| | PPD | |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.

## 1. TABLE OF CONTENTS 6 MILESTONES 12 8. RESEARCH QUESTION AND OBJECTIVES \_\_\_\_\_\_\_\_13 9.2.2 Exclusion Criteria 15 9.4. Data Sources 20 9.5. Study Size 21 9.7. Data Analysis 23 9 9 Limitations of the Research Methods 25 10.2. Patient Consent 26 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS......26 13 REFERENCES 27

| 15. LIST OF FIGURES | 29 |
|---|---|
| 16. APPENDIX | 29 |
| Table 1. Diagnosis Codes for Identifying HIV infection | 29 |
| Table 2. National Drug Codes for Identifying HIV Antiretrovirals (see excel) | 29 |
| Table 3. National Drug Codes and CPT® Codes for Identifying PCV13 Vaccination | n .29 |
| Table 5. Diagnosis Codes for Identifying Pneumococcal Pneumonia and Pneumonium Unspecified Causes | |
| Table 4. Diagnosis Codes for Identifying Invasive Pneumococcal Disease, All-Cau<br>Pneumonia, and Pneumococcal Pneumonia | |
| Table 6. National Drug Codes and Procedure Codes for Identifying Immunosuppre<br>Medications (see excel) | |
| Table 7. National Drug Codes and Procedure Codes for Identifying Influenza Vaccinations (see excel) | 41 |
| Table 8. National Drug Codes and CPT® Codes for Identifying PPSV23 Vaccination | on41 |
| Table 9. CPT® codes to identify CD4 laboratory tests | 42 |
| Table 10. CPT® codes to identify viral load laboratory tests | 42 |
| Table 11. Diagnosis Codes for Identifying All-Cause Pneumonia not due to HIV | 43 |
| Table 12. National Drug Codes and CPT® Codes for Identifying Recombinant Zos<br>Vaccination | |
| Table 13. National Drug Codes for Identifying Candidiasis Antifungals (see excel) | 46 |
| Table 14. Diagnosis Codes for Identifying Opportunistic Infections (see excel) | 46 |
| ANNEX 1. LIST OF STAND ALONE DOCUMENTS | 46 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS | 46 |
| ANNEY 2 ADDITIONAL INCOPMATION | 16 |

## 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| ART | Antiretroviral therapy |
| CAP | Community-acquired pneumonia |
| CAPiTA | The Community-Acquired Pneumonia Immunization<br>Trial in Adults |
| CI | Confidence interval |
| CIOMS | Council for International Organizations of Medical<br>Sciences |
| CPT | Current procedural terminology® |
| CSF | Cerebrospinal fluid |
| EC | Ethics Committee |
| EMA | European Medicines Agency |
| ENCePP | European Network of Centres for<br>Pharmacoepidemiology and Pharmacovigilance |
| FDA | Food and Drug Administration |
| GEP | Good Epidemiological Practice |
| GPP | Good Pharmacoepidemiology Practices |
| HCPCS | Healthcare Common Procedure Coding System |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human immunodeficiency virus |
| HR | Hazard ratio |
| ICD-9-CM | International Classification of Diseases, Ninth Revision,<br>Clinical Modification |

| Abbreviation | Definition |
|---|---|
| ICD-10-CM | International Classification of Diseases, Tenth Revision,<br>Clinical Modification |
| ICD-9-PCS | International Classification of Diseases, Ninth Revision,<br>Procedure Coding System |
| ICD-10-PCS | International Classification of Diseases, Tenth Revision,<br>Procedure Coding System |
| IEA | International Epidemiological Association |
| IPD | Invasive pneumococcal disease |
| IRB | Institutional review board |
| ISPOR | International Society for Pharmacoeconomics and<br>Outcomes Research |
| NDC | National Drug Code |
| PCV | Pneumococcal conjugate vaccine |
| PCV13 | 13-valent pneumococcal conjugate vaccine |
| PCV15 | 15-valent pneumococcal conjugate vaccine |
| PCV20 | 20-valent pneumococcal conjugate vaccine |
| PPSV23 | 23-valent pneumococcal polysaccharide vaccine |
| PLWH | People living with HIV |
| RZV | Recombinant zoster vaccine |
| SVI | Social Vulnerability Index |
| VE | Vaccine effectiveness |
| VT | Vaccine-type |

## 3. RESPONSIBLE PARTIES

Principal Investigator(s) of the Protocol

| Name, Degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| PPD ,<br>PharmD | PPD , US | Pfizer, Inc | 500 Arcola Road<br>Collegeville, PA<br>19426 |

## 4. ABSTRACT

| Title | Assessment of PCV13 vaccine effectiveness among people with HIV |
|---|---|
| Rationale and<br>background | People living with HIV (PLWH) are at increased risk of pneumococcal infections. A recent meta-analysis shows that in the era of advanced antiretroviral therapy, the incidence of invasive pneumococcal disease (IP in PLWH is approximately 30 times higher when compared with the generopopulation [1]. Even with timely and effective treatment, the case fatality rate of IPD is at least 8% in PLWH [2] and up to 25% of PLWH experience recurrent episodes of IPD in the subsequent 12 months [3]. International guidelines recommend pneumococcal vaccination for immunocompromised individuals [4] and previous research has shown that the pneumococcal conjugate vaccine (PCV) is safe and immunogenic in PLWH [5-8]. Studies have assessed the clinical efficacy/effectiveness of PCV in adults, but patients with immunocompromising conditions or treatments were either excluded from the studies, or vaccine effectiveness (VE) estimates were calculated overall and not specifically among PLWH among people with other immunocompromising conditions [9, 10]. |
| | Given the lack of PCV13 VE data in immunocompromised adults, this study was designed to estimate PCV13 VE against pneumococcal disease in PLWH aged ≥18 years, overall and, if feasible, at 3, 5, and 7 years after vaccination. |
| Research | The primary objectives include: |
| objectives | Estimate vaccine effectiveness (VE) of PCV13 for invasive pneumococcal disease (IPD) among people living with HIV (PLWH) ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up |
| | <ol> <li>Estimate VE of PCV13 for pneumococcal pneumonia among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up</li> </ol> |
| | 3. Estimate VE of PCV13 for all-cause pneumonia among PLWH≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up |
| | The secondary objectives of this study are to: |
| | <ol> <li>Estimate VE of PCV13 for pneumococcal pneumonia or pneumonia<br/>with unspecified causes among PLWH ≥18 years of age, overall and,<br/>if feasible, at 3, 5, and 7 years of follow-up</li> </ol> |

| | <ol> <li>Estimate VE of PCV13 for pneumonia with unspecified causes<br/>among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7<br/>years of follow-up</li> </ol> |
|---|---|
| Design | The VE study will be a retrospective cohort study using health care administrative claims and laboratory data. |
| Population | PLWH will be identified using administrative claims and include individuals with at least one inpatient International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code related to HIV or at least 2 outpatient ICD-9-CM or ICD-10-CM codes related to HIV at least 30 days, but no more than 730 days apart, during January 1, 2014 and December 31, 2021. PLWH are required to have at least six months of continuous enrollment in one or more health plans and pharmacy benefits after their first HIV-related ICD-9-CM or ICD-10-CM. These six months of continuous enrollment will be considered the baseline period, during which baseline covariates including demographics, comorbidities, and preventative care will be measured. The end of the study will occur on the last date that administrative claims data will be available, September 30, 2022. |
| Data source | Health care administrative claims and laboratory data will be provided by Komodo Health. Komodo Health uses artificial intelligence and data analytics to combine and link patient-level information from more than 150 payers in the United States, including Medicare, Medicaid, and Commercial plans. Currently, Komodo Health has patient-level data on approximately 325 million individuals and these data include inpatient and outpatient claims, pharmacy dispensing claims, provider specialty claims, and mortality information. |
| Data analyses | Cox proportional hazards models will be used to estimate the hazard ratio (HR) for each outcome comparing vaccinated PLWH with unvaccinated (no PCV13) PLWH. To explore potential changes in VE over time, HRs will also be generated during specific time periods (0-3, 3-5, 5-7 years) using piecewise Cox regression models, if there is adequate sample size. All models will be adjusted for time-fixed and time-varying covariates of interest using inverse probability of treatment weighting. VE will be calculated as 1 minus the estimated HR for each outcome. |

## 5. AMENDMENTS AND UPDATES

| Version | Date | Amendment | Protocol | Summary of | Reason |
|---|---|---|---|---|---|
| Identifier | Date | Type<br>(substantial or<br>administrative) | Section(s)<br>Changed | Amendment(s) | Avenous |
| 2.0 | 02 August 2023 | Substantial | 9.1 Study Design | Individuals must now have at least one inpatient or at least two outpatient HIV-related ICD-9-CM and ICD-10-CM codes occurring at least 30 days but no more than 730 days apart Study follow-up will now begin 90 days after index date | 1. Limiting the time between outpatient HIV diagnosis codes decreases misclassification of HIV infection in administrative claims data 2. Starting follow-up 90 days after index decreases the likelihood that outcome events occurred before and/or triggered an HIV diagnosis |
| | | | 9.3 Variables | 1. Added time-varying covariate for annual HIV viral load testing 2. Added time-varying covariate for annual CD4 cell count testing 3. Added time-varying covariate for respiratory virus season 4. Added an alternate definition for outpatient candidiasis infection (ICD-9-CM or ICD-10-CM code and antifungal treatment within 7 days 5. Changed payor categories | 1. Minimize confounding due to different HIV care seeking patterns among PCV13 vaccinated and unvaccinated individuals 2. Minimize confounding due to different HIV care seeking patterns among PCV13 vaccinated and unvaccinated individuals 3. Minimize confounding due to increased risk for respiratory virus infections during fall and winter months 4. Increase specificity of candidiasis infections within administrative claims 5. Revised payor categories match actual payor categories in data provided by Komodo |
| | | | 9.5 Study size | Added 'Total number of<br>events' columns to Tables 2<br>and 3 | Demonstrates that the study has<br>sufficient statistical power for<br>IPD and all-cause pneumonia<br>outcomes |
| | | | 9.7 Data analysis | Restricted stratified analysis<br>by index year to first 3 years<br>of follow-up | Due to possible waning of the VE and different lengths of follow-up by index year, VE stratification by year of HIV diagnosis will be restricted to the first 3 years of follow-up. |
| | | | Appendix | Added Appendix Table for CD4 cell count laboratory CPT codes | Added Appendix Table 9, 10, and<br>13 as new variables are now<br>included |

| | | | | Added Appendix Table 10 for HIV viral load laboratory CPT codes Added Appendix Table 13 for candidiasis antifungal NDCs | |
|---|---|---|---|---|---|
| 3.0 | 21 November<br>2023 | Substantial | 9.1 Study Design | 1. Removed requirement for six months of continuous enrollment before members' first HIV-related ICD-9-CM or ICD-10-CM code 2. Study follow-up begins six months after the first HIV-related ICD-9-CM or ICD-10-CM code | Analysis will include incident and<br>prevalent HIV cases during 2014 -<br>2021, rather than only including<br>incident cases during 2015-2021 |
| | | | 9.2.1 Inclusion<br>criteria | 1. Removed criterion for six months of continuous enrollment before first HIV-related ICD-9-CM or ICD-10-CM code 2. Require at least six months of continuous enrollment after the first HIV-related ICD-9-CM or ICD-10-CM code instead of 90 days. | Analysis will include incident and<br>prevalent HIV cases during 2014 -<br>2021, rather than only including<br>incident cases during 2015-2021 |
| | | | 9.2.2 Exclusion<br>criteria | Removed exclusion for<br>individuals with evidence of<br>ART therapy during<br>baseline period | Analysis will include incident and<br>prevalent HIV cases during 2014 -<br>2021, rather than only including<br>incident cases during 2015-2021 |
| | | | 9.3 Variables | Added additional opportunistic infections to covariates measured during baseline and follow-up Removed specific negative control exposure and negative control outcomes from table | Control for potential confounding due to any opportunistic infection Study team would like to explore additional negative control exposures and outcomes in analyses beyond Shingrix and candidiasis |
| | | | Appendix | Added additional ICD-9-<br>CM and ICD-10-CM codes<br>for opportunistic infections | Provided diagnosis codes to<br>identify additional opportunistic<br>infections |

#### 6. MILESTONES

| Milestone | Planned date |
|--------------------------|-----------------|
| Start of data collection | 06 March 2023 |
| End of data collection | 30 October 2024 |
| Final study report | 30 October 2024 |

#### 7. RATIONALE AND BACKGROUND

Human immunodeficiency virus (HIV) infection leads to extensive defects in the immune system, including the progressive depletion and dysfunction of CD4<sup>+</sup> T cells, perturbation of the B cell compartment with reduced resting memory B cells, and suboptimal humoral immune responses [11-14]. People living with HIV (PLWH) are at increased risk of pneumococcal infections. While antiretroviral therapy (ART) can restore the immune system and consequently lower the risk of pneumococcal infections [2, 15], the burden of pneumococcal infections persists in PLWH [16, 17]. A recent meta-analysis shows that in the era of advanced ART, the incidence rate of invasive pneumococcal disease (IPD) in PLWH is approximately 30 times higher when compared with the general population [1]. Even with timely and effective treatment, the case fatality rate of IPD is at least 8% in PLWH [2]. Up to 25% of PLWH experience recurrent episodes of IPD in the subsequent 12 months [3].

International guidelines recommend pneumococcal vaccination for immunocompromised individuals [4]. In the United States, one dose of 13-valent pneumococcal conjugate vaccine (PCV13) has been recommended to PLWH since 2012 [18]. Currently, the CDC recommends 20-valent pneumococcal conjugate vaccine (PCV20) alone or 15-valent pneumococcal conjugate vaccine (PCV15) followed by pneumococcal polysaccharide vaccine (PPSV23) for adults aged 19-64 years with certain underlying medical conditions, including HIV infection, and for all adults aged ≥65 years [19].

Previous research has shown that PCV13 is safe and immunogenic in adults, including PLWH [5-8]. A few studies also assessed the clinical efficacy/effectiveness of a PCV in adults. In a large, randomized, placebo-controlled clinical trial (CAPiTA) of over 84,000 Dutch adults aged ≥65 years, PCV13 showed efficacy against both vaccine-type (VT) IPD (VE 75%; 95% confidence interval [CI]: 41% to 91%) and VT non-bacteremic pneumococcal community-acquired pneumonia (CAP) (VE 45%; 95 % CI: 14%-65%) [9]. PCV13 efficacy persisted throughout the clinical trial (mean follow-up: 4 years) [9]. A population-based, test negative design, surveillance study reported a PCV13 VE of 73% (95% CI: 13%-92%) against VT CAP in hospitalized adults aged ≥65 years [10]. In a clinical trial conducted in HIV-infected adults in Malawi recently hospitalized with pneumonia, two doses of PCV7 demonstrated substantial protection against recurrent pneumococcal infection caused by vaccine serotypes or serotype 6A (VE 74%; 95% CI: 30%-90%) [3], although there was no protection against mortality.

Although the CAPiTA study provides important information on PCV13 VE in adults, patients with any immunocompromising condition or treatment were excluded from the study. In contrast to CAPiTA, the study by McLaughlin et al. included immunocompromised adults; however, PCV13 VE was reported for the entire study population [10]. Thus, there is a lack of data on PCV13 VE specific to immunocompromised adults. In the absence of such data, in a CDC cost-effectiveness PFIZER CONFIDENTIAL

model, it was assumed that PCV13 VE in immunocompromised adults was 25% (95% CI: 14%-30%) against VT IPD and 15% (95% CI: 5%-22%) against VT pneumonia, both of which are approximately one third of the VE measured in healthy adults/adults with chronic medical conditions [20, 21].

There has been a longstanding recommendation for pneumococcal vaccination for PLWH in the United States. PCV13 was recommended for PLWH in 2012 and the uptake in PLWH is higher compared with individuals with other risk conditions [22, 23]; this allows us to examine PCV13 VE in the PLWH population over time. Given the lack of PCV13 VE data in immunocompromised adults, this study was designed to estimate PCV13 VE against pneumococcal disease in PLWH aged ≥18 years, overall and, if feasible, at 3, 5, and 7 years after vaccination. In addition to IPD and pneumococcal pneumonia, we will include all-cause pneumonia as a disease endpoint in the analysis, because *S. pneumoniae* is the most common bacterial cause of all-cause pneumonia [24].

## 8. RESEARCH QUESTION AND OBJECTIVES

The primary objectives of this study are:

- Estimate VE of PCV13 for IPD among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- Estimate VE of PCV13 for pneumococcal pneumonia among PLWH≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- Estimate VE of PCV13 for all-cause pneumonia among PLWH≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up

The secondary objectives of this study are:

- Estimate VE of PCV13 for pneumococcal pneumonia or pneumonia with unspecified causes among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- Estimate VE of PCV13 for pneumonia with unspecified causes among PLWH ≥18
  years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up

#### 9. RESEARCH METHODS

## 9.1. Study Design

The VE study will be a retrospective cohort study using health care administrative claims and laboratory data (Figure 1).

PLWH will be identified using administrative claims and include individuals with at least one inpatient International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code related to HIV (Appendix Table 1) or at least 2 outpatient ICD-9-CM or ICD-10-CM codes related to HIV at least 30 days, but no more than 730 days apart, during January 1, 2014 and

December 31, 2021. PLWH are required to have at least six months of continuous enrollment in one or more health plans and pharmacy benefits after their first HIV-related ICD-9-CM or ICD-10-CM code. These six months of continuous enrollment will be considered the baseline period, during which baseline covariates including demographics, comorbidities, and preventative care will be measured. The baseline period was also selected to minimize the number of outcome events that existing prior to or triggered an HIV diagnosis.

The date following the last date of the baseline period will be defined as the index date. The end of the study will occur on the last date that administrative claims data will be available, September 30, 2022.

For PLWH who receive PCV13 after their index date, we will include the time between their index date and the 13 days after their PCV13 vaccination date as unvaccinated follow-up time. Any outcomes occurring during this time will be counted as events in the unvaccinated cohort. Follow-up that occurs 14 days or more after PCV13 vaccination will be defined as vaccinated follow-up time.

Unvaccinated (no PCV13) PLWH will be followed from index date until the earliest occurrence of the following: 13 days after PCV13 vaccination, death, end of health plan enrollment, or end of study period. Vaccinated PLWH will be followed from 14 days after their PCV13 vaccination, or index date if they were vaccinated during the baseline period, until the earliest occurrence of the following: death, end of health plan enrollment, or end of study period.

### 9.2. Setting

Health care administrative claims and laboratory data will be provided by Komodo Health. Komodo Health uses artificial intelligence and data analytics to combine and link patient-level information from more than 150 payers in the United States, including Medicare, Medicaid, and Commercial plans.

Komodo Health will provide administrative claims data and HIV-related laboratory data available during January 1, 2014 through September 30, 2022 for individuals who have at least one ICD-9-CM or ICD-10-CM code related to HIV (Appendix Table 1) or at least one ART medication dispensed (Appendix Table 2).

## 9.2.1. Inclusion Criteria

To be eligible for the vaccine effectiveness study, individuals must meet the following criteria:

 HIV infection defined as at least one inpatient International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code related to HIV (Appendix Table 1) or ≥2 outpatient ICD-9-CM or ICD-10-CM codes related to HIV at least 30 days, but no more than 730 days apart, during January 1, 2014 and December 31, 2021

AND

At least 18 years of age at the time of the first recording of HIV-related ICD-9-CM or ICD-10-CM code

AND

 At least six months of continuous enrollment in medical and pharmacy plans after the first HIV-related ICD-9-CM or ICD-10-CM code between January 1, 2014 and December 31, 2021. A gap of 30 days or less in enrollment will be allowed during this six month period.

#### 9.2.2. Exclusion Criteria

Patients meeting the following criterion will not be included in the study:

1. Evidence of PCV13 vaccination before the first HIV-related ICD-9-CM or ICD-10-CM code

Figure 1. Illustrative timeline for study participants



## 9.3. Variables

Table 1. Variables, definitions, and measurement periods

| Variable<br>type | Variable | Definition | Measurement<br>period |
|---|---|---|---|
| Exposure | PCV13 vaccination | Current procedural<br>terminology® (CPT) codes and<br>National Drug Codes (NDC)<br>listed in Appendix Table 3 | Follow-up |
| Primary<br>outcomes | IPD | ICD-9-CM or ICD-10-CM codes<br>listed in Appendix Table 4 | Follow-up |
| | Pneumococcal<br>pneumonia | ICD-9-CM or ICD-10-CM codes<br>listed in Appendix Table 4 | Follow-up |
| | All-cause pneumonia | ICD-9-CM or ICD-10-CM codes<br>listed in Appendix Table 4 | Follow-up |
| | Pneumococcal<br>pneumonia or<br>pneumonia with<br>unspecified causes | ICD-9-CM or ICD-10-CM codes<br>listed in Appendix Table 5 | Follow-up |
| | Pneumonia with<br>unspecified causes | ICD-9-CM or ICD-10-CM codes<br>listed in Appendix Table 5 | Follow-up |
| Covariates | Age | Calculated as [year individual meets HIV criteria] – [birth year] Categorized as 18-49, 50-64, 65-74, and ≥75 years | Baseline |
| | Sex | Male, Female, Other, Unknown | Baseline |
| | Social Vulnerability<br>Index (SVI) | SVI characterizes resiliency of a community when faced by external pressures and stresses [25, 26]. SVI ranges from 0 to 100, where a value of 100 indicates the most vulnerable population. SVI will be estimated using zip code and will be categorized as low (lowest quartile), average (middle two quartiles) and high (highest quartile). | Baseline |
| | Payor | yor Medicaid/CHIP, Medicare,<br>Commercial, Dually eligible,<br>Other, Unknown | |
| | US region | Northeast, North Central, South,<br>West, Unknown | Baseline |

| Variable<br>type | Variable | Definition | Measurement<br>period |
|---|---|---|---|
| | Index year | Calendar year of first HIV diagnosis code | Baseline |
| | Alcoholism | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.1 | follow-up |
| | Asplenia | CPT/Healthcare Common | Baseline and |
| | | Procedure Coding System | follow-up |
| | | (HCPCS), ICD-10-Procedure | |
| | | Coding System (ICD-10-PCS), | |
| | | ICD-9-Procedure Coding System | |
| | | (ICD-9-PCS), ICD-9-CM, or | |
| | | ICD-10-CM codes listed in | |
| | | Annex Table 1.2 | |
| | Asthma | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.3 | follow-up |
| | Chronic heart disease | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | | ICD-9-PCS, ICD-9-CM, or ICD- | follow-up |
| | | 10-CM codes listed in Annex | |
| | | Table 1.4 | |
| | Chronic kidney | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | disease and renal | ICD-9-PCS, ICD-9-CM, or ICD- | follow-up |
| | failure | 10-CM codes listed in Annex | |
| | | Table 1.5 | |
| | Chronic liver disease | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | | ICD-9-PCS, ICD-9-CM, or ICD- | follow-up |
| | | 10-CM codes listed in Annex | |
| | | Table 1.6 | |
| | Chronic lung disease | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.7 | follow-up |
| | Cigarette smoking | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.8 | follow-up |
| | Diabetes mellitus | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.9 | follow-up |
| | Generalized | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | malignancy | ICD-9-PCS, ICD-9-CM or ICD- | follow-up |
| | | 10-CM codes listed in Annex | |
| | TT- 4-1-i-2- 11 - | Table 1.10 | Danalius and |
| | Hodgkin's lymphoma | ICD-9-CM or ICD-10-CM codes<br>listed in Annex Table 1.11 | Baseline and follow-up |
| | Immunosuppressive | PLWH will considered on | Baseline and |
| | medications | immunosuppressive medications | follow-up |
| | | if: | |

| Variable | Variable | Definition | Measurement |
|---|---|---|---|
| type | | | period |
| | | 1)≥1 NDC, HCPCS, or ICD-10- | |
| | | PCS code in Appendix Table 6 | |
| | | 2) $\geq$ 1 NDC (using orals only) in | |
| | | Appendix Table 6 where the | |
| | | daily dose is $\geq$ 20mg or | |
| | | prednisone or prednisone | |
| | | equivalent for a duration of ≥14 | |
| | | consecutive days | |
| | Leukemia | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.12 | follow-up |
| | Multiple myeloma | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.13 | follow-up |
| | Nephrotic syndrome | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 1.14 | follow-up |
| | Non-Hodgkin's | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | lymphoma | listed in Annex Table 1.15 | follow-up |
| | Organ transplant | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | | ICD-9-PCS, ICD-9-CM or ICD- | follow-up |
| | | 10-CM codes listed in Annex | _ |
| | | Table 1.16 | |
| | Sickle cell disease or | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | other | listed in Annex Table 1.17 | follow-up |
| | hemoglobinopathies | | _ |
| | Hepatitis B | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | | listed in Annex Table 2.1 | follow-up |
| | Hepatitis C | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | _ | listed in Annex Table 2.2 | follow-up |
| | Annual physical exam | CPT/HCPCS codes listed in | Baseline and |
| | | Annex Table 3.1 | follow-up |
| | Annual influenza | CPT/HCPCS, ICD-10-PCS, | Baseline and |
| | vaccine | ICD-9-PCS, or NDC codes listed | follow-up |
| | | in Appendix Table 7 | |
| | Any pneumonia | ICD-9-CM or ICD-10-CM codes | Baseline |
| | infection | listed in Appendix Table 4 | |
| | Any hospitalization | Evidence of inpatient claims | Baseline and |
| | ' ' | <b>,</b> | follow-up |
| | Opportunistic | ICD-9-CM or ICD-10-CM codes | Baseline and |
| | infections | listed in Appendix Table 14 | follow-up |
| | ART adherence | ART use will be identified by | Baseline and |
| | | NDC codes listed in Appendix | follow-up |
| | | Table 2 | • |

| Variable | Variable | Definition | Measurement |
|---|---|---|---|
| type | | | period |
| | | Adherence will be measured as | |
| | | 'Proportion of days covered = | |
| | | (Number of days covered by any | |
| | | ART, excluding ritonavir and | |
| | | cobicistat) ÷ (total | |
| | | days)*100'[27] every six months | |
| | | Individuals with >80% of days | |
| | | covered will be classified as | |
| | | 'adherent' and individuals with | |
| | | ≤80% of days covered will be | |
| | | classified as 'non-adherent' [27] | |
| | CD4 cell count | Categorized as <200, 200-499, | Baseline and |
| | | ≥500 cells/mm³ | follow-up |
| | PPSV23 vaccination | NDC and CPT codes listed in | Baseline and |
| | | Appendix Table 8 | follow-up |
| | Annual CD4 | CD4 laboratory tests will be | Baseline and |
| | laboratory test | identified by CPT codes listed in | follow-up |
| | , | Appendix Table 9 | • |
| | | Individuals who have at least | |
| | | one CD4 laboratory test | |
| | | performed during each year of | |
| | | follow-up | |
| | Annual viral load | Viral load laboratory tests will | Baseline and |
| | laboratory test | be identified by CPT codes listed | follow-up |
| | | in Appendix Table 10 | • |
| | | Individuals who have at least | |
| | | one viral load laboratory test | |
| | | performed during each year of | |
| | | follow-up | |
| | Respiratory virus | Respiratory virus season occurs | Follow-up |
| | season | between October 1 and April 30 | • |
| Sensitivity | All-cause pneumonia | ICD-9-CM or ICD-10-CM codes | Follow-up |
| analysis | not associated with | listed in Appendix Table 11 | • |
| outcome | HIV | | |

## 9.4. Data Sources

The source of data for the VE study will be health care administrative claims and HIVlaboratory data provided by Komodo Health. Komodo Health uses artificial intelligence and

data analytics to combine and link patient-level information from more than 150 payers in the United States, including Medicare, Medicaid, and Commercial plans. Currently, Komodo Health has patient-level data on approximately 325 million individuals and these data include inpatient and outpatient claims, pharmacy dispensing claims, provider specialty claims, and mortality information.

Komodo Health will provide administrative claims available between January 1, 2014 through September 30, 2022 for individuals who have at least one ICD-9-CM or ICD-10-CM code related to HIV (Appendix Table 1) or at least one ART medication dispensed (Appendix Table 2).

### 9.5. Study Size

The planned analyses do not involve hypothesis testing and sample size calculations are not applicable. However, we examined the precision of PCV13 vaccine effectiveness for IPD and all-cause pneumonia among people living with HIV at 36 months and 97 months (which was the maximum follow-up time available from feasibility assessments) after index (Table 2 and Table 3). Komodo Health provided the following information for the precision estimates:

- 175,000 individuals had ≥1 inpatient or ≥ 2 outpatient HIV ICD-9-CM or ICD-10-CM code diagnosis codes between January 1, 2014 and December 31, 2021
- 56,000 (32%) of these individuals received PCV13 after their first HIV diagnosis code

The following assumptions regarding incidence and PCV13 VE for IPD and all-cause pneumonia were used:

- IPD incidence among PLWH is 183 cases per 100,000 population [28]
- All-cause pneumonia incidence among PLWH is 5,487 cases per 100,000 population
- VE for IPD due to any serotype ranges from 7.5% to 22.5%
  - Published VE estimates for vaccine type IPD range from 25% to 75% [20].
     Because one-third of the adult IPD burden is considered PCV13 type [29], we multiplied this range by 30% to arrive at 7.5% to 22.5%
- VE for all-cause pneumonia ranges from 5% to 15% [30]
- Annual censoring of individuals due to loss to follow-up or death may range between 4% or 10%

Survival and censoring times were simulated assuming exponential distributions. Vaccination status was modelled as a time-varying covariate [31]. Hazard ratios were assumed as 1 - (VE/100). Simulations were run 100 to 200 times per scenario. Cox regression models were run on each simulated dataset to estimate the 95% confidence PFIZER CONFIDENTIAL

intervals (CI) for the log HRs. Means were generated and exponentiated to obtain the 95% CIs for the VEs using (1 - HR) x 100 and used to describe VE precision.

Table 2. Precision of PCV13 vaccine effectiveness estimates for invasive pneumococcal disease

| Hypothesized | 36 months of follow-up | | | 97 months of follow-up | | ow-up |
|---|---|---|---|---|---|---|
| Vaccine | Lower | Upper | Total | Lower | Upper | Total |
| Effectiveness | 95% | 95% | number of | 95% | 95% | number of |
| (%) | confidenc | confidenc | events | confidenc | confidenc | events |
| | e interval | e interval | | e interval | e interval | |
| | estimate | estimate | | estimate | estimate | |
| Scenario #1 – 49 | % annual cen | soring | | | | |
| 7.5 | -12 | 25 | 837 | -5 | 19 | 1492 |
| 22.5 | 3 | 37 | 817 | 11 | 33 | 1452 |
| Scenario #2 – 10% annual censoring | | | | | | |
| 7.5 | -15 | 25 | 766 | -6 | 21 | 1272 |
| 22.5 | 2 | 38 | 752 | 9 | 33 | 1224 |

Table 3. Precision of PCV13 vaccine effectiveness estimates for all-cause pneumonia

| Hypothesized | 36 months of follow-up | | | 97 months of follow-up | | |
|---|---|---|---|---|---|---|
| Vaccine | Lower | Upper | Total | Lower | Upper | Total |
| Effectiveness | 95% | 95% | number of | 95% | 95% | number of |
| (%) | confidenc | confidenc | events | confidenc | confidenc | events |
| | e interval | e interval | | e interval | e interval | |
| | estimate | estimate | | estimate | estimate | |
| Scenario #1 – 49 | % annual cen | soring | | | | |
| 5 | 1 | 9 | 23,370 | 2 | 7 | 38,848 |
| 15 | 11 | 19 | 23,119 | 13 | 17 | 38,176 |
| Scenario #2 – 10% annual censoring | | | | | | |
| 5 | 1 | 9 | 21,558 | 2 | 8 | 33,257 |
| 15 | 11 | 19 | 21,327 | 12 | 18 | 32,750 |

Given the precision estimates in Tables 1 and 2, the planned study should have adequate precision to address the primary objectives.

## 9.6. Data Management

Komodo will create analytic files comprising people who have at least one HIV related ICD-9-CM or ICD-10-CM code or claim for an ART medication to treat HIV. The analytic files will include person-level data, including information on baseline demographic and clinical characteristics, study outcomes, and health plan enrollment dates. Variables will be created based on information from healthcare claims and enrollment information, which will be

linked at the person level using a unique ID, which is deidentified. Data for this study will be processed and managed by Pfizer, Inc., and all analyses—as described in the final version of the Study Protocol—will be directed by study investigators.

Retention of study-related data, documents, and other materials will be governed by Pfizer Policy on Records and Information Management, and per this policy, will remain effective for a period of 5 years from the date of project initiation. Amendments must be made only with the prior approval of Pfizer. Agreement from all study collaborators must be obtained for all amendments.

#### 9.7. Data Analysis

Cox proportional hazards models will be used to estimate the hazard ratio (HR) for each outcome comparing vaccinated PLWH with unvaccinated (no PCV13) PLWH. To explore potential changes in VE over time, HRs will also be generated during specific time periods (0-3, 3-5, 5-7 years of follow-up) using piecewise Cox regression models, if there is adequate sample size. All models will be adjusted for time-fixed and time-varying covariates of interest using inverse probability of treatment weighting. The time-fixed covariates of interest include sex, age, payor, SVI, previous pneumonia infection, and hospitalization and will be measured during the baseline period. The time-varying covariates include risk factors for pneumonia (alcoholism, asplenia, asthma, chronic heart disease, kidney, liver, and lung diseases, cigarette smoking, diabetes, immunosuppressive conditions and medications, and sickle cell disease), annual physical exams, annual influenza vaccine, hospitalization, opportunistic infections, ART adherence, annual CD4 and viral load laboratory tests, and an indicator for respiratory virus season.

VE will be calculated as 1 minus the estimated HR for each outcome.

We will conduct two sets of analyses for each outcome. In the first set, we will examine the first event for each outcome and in the second set, all recurrent outcome events during follow-up will be included. In the first set of analyses, unvaccinated (no PCV13) PLWH will be followed from index date until the earliest occurrence of the following: outcome, PCV13 vaccination, death, end of health plan enrollment, or end of study period, and vaccinated PLWH will be followed from 14 days after vaccination date, or index date if vaccinated during the baseline period, until the earliest occurrence of outcome, death, end of health plan enrollment, or end of study period. In the second set of analyses unvaccinated (no PCV13) PLWH will be followed from index date until the earliest occurrence of PCV13 vaccination, death, end of health plan enrollment or end of study period and vaccinated PLWH will be followed from 14 days after vaccination date, or index date if vaccinated during the baseline period, until earliest occurrence of death, end of health plan enrollment, or end of study period.

Several stratified analyses will be conducted. PPSV23 is recommended for PLWH and feasibility data provided by Komodo suggest that one in four PWLH who received PCV13 during 2014-2015 also received PPSV23 within two years. Rather than censor or exclude

individuals who receive PPSV23, we will calculate PCV13 VE among PWLH who have/have not received PPSV23 before and during the study period.

Feasibility assessments from Komodo indicate that approximately 25% of PWLH have at least one CD4 cell count or percentage laboratory result available. Therefore, we will calculate PCV13 VE among the subset of PWLH who have a CD4 cell count during the baseline period or follow-up, and potentially stratify by CD4 category using each patient's lowest value during the study.

Additional VE stratifications by ART adherence during follow-up, year of HIV diagnosis, and age will be assessed for feasibility as well, as these affect patients' immune status and immune reconstitution. Due to possible waning of the VE and different lengths of follow-up by index year, VE stratification by year of HIV diagnosis will be restricted to the first 3 years of follow-up.

A sensitivity analysis will also be conducted. In this analysis, causes of pneumonia that are characteristic of HIV, for example pneumonia due to cytomegalovirus, mycobacteria, and fungi, will be excluded from our definition of all-cause pneumonia.

Residual confounding of our VE estimates due to inadequate control for health care seeking behavior and immune status in our analyses will be explored. To do so, we will employ a negative control exposure and a negative control outcome. Potential negative control exposures include vaccinations that are recommended for PLWH but would not be expected to have any protective effect against the pneumonia outcomes of interest. If residual confounding does not exist, the negative control vaccine would not have an effect on the pneumonia outcomes. However, if the analysis demonstrates that the negative control vaccine protects against these outcomes, this suggests the presence of residual confounding.

Similarly, potential negative control outcomes are outcomes that share the same sources of biases as the primary outcomes in our study population but are not causally-related to PCV13 vaccination. For example, immune status is an important predictor of pneumonia outcomes among PLWH, but we will be missing CD4 laboratory values for most of our study population. In order to detect potential residual confounding by lack of control for immune status, a potential negative control outcome could include a more common AIDS defining illness such as candidiasis. Again, if no residual confounding exists, PCV13 vaccination would have no effect on the occurrence of the negative control outcomes. However, if the results suggest that PCV13 vaccination prevents the negative control outcomes, residual confounding may exist.

Detailed methodology for summary and statistical analyses of data collected in this study will be documented in a statistical analysis plan (SAP), which will be dated, filed and maintained by the sponsor. The SAP may modify the plans outlined in the protocol; any major modifications of primary endpoint definitions or their analyses would be reflected in a protocol amendment.

## 9.8. Quality Control

Upon initiation of analyses, edit, range, and logic checks will be performed on each data field by the project programmer to ensure the quality and completeness of the study database and all of the variables therein. Only observed data will be used in measuring study variables. It is anticipated that demographic information will be available for nearly all individuals in the study population. All other variables will be defined based on the presence of specific data (e.g., diagnosis, procedure, and drug codes) in the analytic file; the absence of such data will be assumed to indicate the absence of the characteristic/event captured by the variable.

#### 9.9. Limitations of the Research Methods

There are several limitations in this study. Given that this is an observational study using health care administrative claims data, residual confounding due to missing or unmeasured information is possible. To examine this, we will assess the effect of PCV13 on a negative control outcome and the effect of a negative control exposure on our outcomes of interest. If the HRs in any of these models are less than 1.0, it would indicate that residual confounding exists and may result in adjustment of our VE estimates.

Second, health care administrative claims data will be available from January 1, 2014 through September 30, 2022. The recommendation to vaccinate all PLWH was published in June 2012, and some PLWH may have received PCV13 prior to January 1, 2014 and be misclassified as unvaccinated. In addition, PLWH eligible for the study may have received PCV13 vaccination during a time period in which we do not have their claims data. Misclassification of PCV13 vaccine status may lead to lower estimates of vaccine effectiveness than in truth, because our unvaccinated cohort will incorrectly include vaccinated PLWH.

In addition, we are using ICD-9-CM and ICD-10-CM codes to define HIV infection. Our definition of HIV infection requires at least one HIV-related diagnosis code in the inpatient setting or at least two HIV-related diagnosis codes in the outpatient setting. While this definition of HIV has been used in previous administrative claims database studies, it is possible that these codes may be used by health care providers to order laboratory tests to rule out HIV infection and thus, some individuals without HIV will be included in our study population.

## 9.10. Other Aspects

Not applicable

#### 10. PROTECTION OF HUMAN PARTICIPANTS

#### 10.1. Patient Information

This study involves data that exist in deidentified/anonymized structured format and contain no patient personal information.

#### 10.2. Patient Consent

As this study involves deidentified/anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

#### 10.3. Institutional Review Board (IRB)/Ethics Committee (EC)

The study databases will be de-identified prior to their release to study investigators, as set forth in the corresponding Data Use Agreement. The study databases have been evaluated and certified by an independent third party to be compliant with the Health Insurance Portability and Accountability Act (HIPAA) of 1996 statistical de-identification standards and to satisfy the conditions set forth in Sections 164.514 (a)-(b)1ii of the HIPAA Privacy Rule regarding the determination and documentation of statistically de-identified data. Use of the study databases for health services research is therefore fully compliant with the HIPAA Privacy Rule and federal guidance on Public Welfare and the Protection of Human Subjects (45 Code of Federal Regulations [CFR] 46 §46.101) and IRB approval is not required.

## 10.4. Ethical Conduct of the Study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in *Good Pharmacoepidemiology Practices* (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA), Good Outcomes Research Practices issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR), International Ethical Guidelines for Epidemiological Research issued by the Council for International Organizations of Medical Sciences (CIOMS), European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacoepidemiology, and Food and Drug Administration (FDA) Guidance for Industry: Good Pharmacovigilance and Pharmacoepidemiologic Assessment, and FDA Draft Guidance for Industry and FDA Staff: Best Practices for Conducting and Reporting of Pharmacoepidemiologic Safety Studies Using Electronic Healthcare Data Sets and/or equivalent.

## 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves data that exist as structured data by the time of study start. In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.

## 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

Formal communication of the results of this research will be done by study investigators through peer-reviewed publications. For all publications relating to the Study, Pfizer will comply with recognized ethical standards concerning publications and authorship, including

Section II - "Ethical Considerations in the Conduct and Reporting of Research" of the Uniform Requirements for Manuscripts Submitted to Biomedical Journals, http://www.icmje.org/index.html#authorship, established by the International Committee of Medical Journal Editors.

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable competent authority in any area of the world, or if the investigator is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

#### 13. REFERENCES

- van Aalst M, Lotsch F, Spijker R, et al. Incidence of invasive pneumococcal disease in immunocompromised patients: A systematic review and meta-analysis. Travel Med Infect Dis 2018; 24: 89-100.
- Grau I, Pallares R, Tubau F, et al. Epidemiologic changes in bacteremic pneumococcal disease in patients with human immunodeficiency virus in the era of highly active antiretroviral therapy. Arch Intern Med 2005; 165(13): 1533-40.
- French N, Gordon SB, Mwalukomo T, et al. A trial of a 7-valent pneumococcal conjugate vaccine in HIV-infected adults. N Engl J Med 2010; 362(9): 812-22.
- Lopez A, Mariette X, Bachelez H, et al. Vaccination recommendations for the adult immunosuppressed patient: A systematic review and comprehensive field synopsis. J Autoimmun 2017; 80: 10-27.
- Bhorat AE, Madhi SA, Laudat F, et al. Immunogenicity and safety of the 13-valent pneumococcal conjugate vaccine in HIV-infected individuals naive to pneumococcal vaccination. AIDS 2015; 29(11): 1345-54.
- Cheng A, Chang SY, Tsai MS, et al. Long-term immune responses and comparative effectiveness of one or two doses of 7-valent pneumococcal conjugate vaccine (PCV7) in HIV-positive adults in the era of combination antiretroviral therapy. J Int AIDS Soc 2016; 19(1): 20631.
- Glesby MJ, Watson W, Brinson C, et al. Immunogenicity and Safety of 13-Valent Pneumococcal Conjugate Vaccine in HIV-Infected Adults Previously Vaccinated With Pneumococcal Polysaccharide Vaccine. The Journal of Infectious Diseases 2014; 212(1): 18-27.
- Sogaard OS, Lohse N, Harboe ZB, et al. Improving the immunogenicity of pneumococcal conjugate vaccine in HIV-infected adults with a toll-like receptor 9 agonist adjuvant: a randomized, controlled trial. Clin Infect Dis 2010; 51(1): 42-50.
- Bonten MJ, Huijts SM, Bolkenbaas M, et al. Polysaccharide conjugate vaccine against pneumococcal pneumonia in adults. N Engl J Med 2015; 372(12): 1114-25.
- McLaughlin JM, Jiang Q, Isturiz RE, et al. Effectiveness of 13-Valent Pneumococcal Conjugate Vaccine Against Hospitalization for Community-Acquired Pneumonia in Older US Adults: A Test-Negative Design. Clinical Infectious Diseases 2018; 67(10): 1498-506.
- Amu S, Ruffin N, Rethi B, Chiodi F. Impairment of B-cell functions during HIV-1 infection. AIDS 2013; 27(15): 2323-34.

- Lee K-Y, Tsai M-S, Kuo K-C, et al. Pneumococcal vaccination among HIV-infected adult patients in the era of combination antiretroviral therapy. Human Vaccines & Immunotherapeutics 2014; 10(12): 3700-10.
- Moir S, Fauci AS. B cells in HIV infection and disease. Nat Rev Immunol 2009; 9(4): 235-45.
- Titanji K, De Milito A, Cagigi A, et al. Loss of memory B cells impairs maintenance of long-term serologic memory during HIV-1 infection. Blood 2006; 108(5): 1580-7.
- Yin Z, Rice BD, Waight P, et al. Invasive pneumococcal disease among HIV-positive individuals, 2000-2009. AIDS 2012; 26(1): 87-94.
- Garcia Garrido HM, Mak AMR, Wit F, et al. Incidence and Risk Factors for Invasive Pneumococcal Disease and Community-acquired Pneumonia in Human Immunodeficiency Virus-Infected Individuals in a High-income Setting. Clin Infect Dis 2020; 71(1): 41-50.
- Sogaard OS, Lohse N, Gerstoft J, et al. Hospitalization for pneumonia among individuals with and without HIV infection, 1995-2007: a Danish population-based, nationwide cohort study. Clin Infect Dis 2008; 47(10): 1345-53.
- CDC. Use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal
  polysaccharide vaccine for adults with immunocompromising conditions:
  recommendations of the Advisory Committee on Immunization Practices (ACIP).
  MMWR Morb Mortal Wkly Rep 2012; 61(40): 816-9.
- Kobayashi M, Farrar JL, Gierke R, et al. Use of 15-Valent Pneumococcal Conjugate Vaccine and 20-Valent Pneumococcal Conjugate Vaccine Among U.S. Adults: Updated Recommendations of the Advisory Committee on Immunization Practices -United States, 2022. MMWR Morb Mortal Wkly Rep 2022; 71(4): 109-17.
- Andrew Leidner. Summary of economic models assessing pneumococcal vaccines in US adults. ACIP Presentation Slides: September 29, 2021 Meeting. Available at: https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2021-09-29/02-Pneumococcal-Leidner-508.pdf. Accessed October 2, 2022.
- Cho BH, Stoecker C, Link-Gelles R, Moore MR. Cost-effectiveness of administering 13-valent pneumococcal conjugate vaccine in addition to 23-valent pneumococcal polysaccharide vaccine to adults with immunocompromising conditions. Vaccine 2013; 31(50): 6011-21.
- Morga A, Kimura T, Feng Q, Rozario N, Schwartz J. Compliance to Advisory Committee on Immunization Practices recommendations for pneumococcal vaccination. Vaccine 2022; 40(15): 2274-81.
- Vietri J, Harnett J, Emir B, Chilson E. Uptake of 13-Valent Pneumococcal Conjugate Vaccine among US Adults Aged 19 to 64 Years with Immunocompromising Conditions. Hum Vaccin Immunother 2020; 16(1): 161-8.
- Said MA, Johnson HL, Nonyane BA, et al. Estimating the burden of pneumococcal pneumonia among adults: a systematic review and meta-analysis of diagnostic techniques. PLoS One 2013; 8(4): e60273.
- CDC's Social Vulnerability Index (SVI). Available at: https://www.atsdr.cdc.gov/placeandhealth/svi/index.html. Accessed November 30, 2022.

- Hyer JM, Tsilimigras DI, Diaz A, et al. High Social Vulnerability and "Textbook Outcomes" after Cancer Operation. J Am Coll Surg 2021; 232(4): 351-9.
- de Oliveira Costa J, Zhao Y, Pearson SA, Schaffer AL. Assessing the impact of implementing multiple adherence measures to antiretroviral therapy from dispensing data: a short report. AIDS Care 2022: 1-6.
- Kobayashi M, Matanock A, Xing W, et al. Impact of 13-Valent Pneumococcal Conjugate Vaccine on Invasive Pneumococcal Disease Among Adults With HIV-United States, 2008-2018. J Acquir Immune Defic Syndr 2022; 90(1): 6-14.
- Ryan Gierke. Current Epidemiology of Pneumococcal Disease, United States-2019 updates. ACIP Presentation Slides: June 25, 2021 Meeting. Available at: https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2021-06/02-Pneumococcal-Gierke-508.pdf. Accessed January 24, 2023.
- Hsiao A, Hansen J, Timbol J, et al. Incidence and Estimated Vaccine Effectiveness Against Hospitalizations for All-Cause Pneumonia Among Older US Adults Who Were Vaccinated and Not Vaccinated With 13-Valent Pneumococcal Conjugate Vaccine. JAMA Netw Open 2022; 5(3): e221111.
- Austin PC. Generating survival times to simulate Cox proportional hazards models with time-varying covariates. Stat Med 2012; 31(29): 3946-58.

#### 14. LIST OF TABLES

| Table 1. Variables, definitions, and measurement periods | 17 |
|---|---|
| Table 2. Precision of PCV13 vaccine effectiveness estimates for invasive pneumococcal disease | 22 |
| Table 3. Precision of PCV13 vaccine effectiveness estimates for all-cause pneumonia | 22 |
| 15. LIST OF FIGURES | |
| Figure 1. Illustrative timeline for study participants | 16 |
| 16. APPENDIX | |

#### Table 1. Diagnosis Codes for Identifying HIV infection

| Code | Type | Description |
|------|-----------|--------------------------|
| 042 | ICD-9-CM | HIV-1 infection |
| V08 | ICD-9-CM | Asymptomatic HIV disease |
| B20 | ICD-10-CM | HIV-1 infection |
| Z21 | ICD-10-CM | Asymptomatic HIV disease |

Table 2. National Drug Codes for Identifying HIV Antiretrovirals (see excel)

## Table 3. National Drug Codes and CPT® Codes for Identifying PCV13 Vaccination

| Code | Type | Description |
|-------------|------|------------------------------------------|
| 50090194409 | NDC | 13-valent pneumococcal conjugate vaccine |
| 54569661300 | NDC | 13-valent pneumococcal conjugate vaccine |

| 50090194400 | NDC | 13-valent pneumococcal |
|-------------|-----|------------------------|
| 30090194400 | NDC | |
| | | conjugate vaccine |
| 00005197105 | NDC | 13-valent pneumococcal |
| | | conjugate vaccine |
| 00005197104 | NDC | 13-valent pneumococcal |
| | | conjugate vaccine |
| 00005197102 | NDC | 13-valent pneumococcal |
| | | conjugate vaccine |
| 00005197101 | NDC | 13-valent pneumococcal |
| | | conjugate vaccine |
| 90670 | CPT | 13-valent pneumococcal |
| | | conjugate vaccine |

Table 5. Diagnosis Codes for Identifying Pneumococcal Pneumonia and Pneumonia with Unspecified Causes

| | | ICD-9-CM | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| | 481 | Pneumococcal pneumonia | J13 | Pneumonia due to Streptococcus pneumoniae |
| | 482.9 +<br>041.2 | Bacterial pneumonia,<br>unspecified + pneumococcus | J15.9 + B95.3 | Unspecified bacterial pneumonia + Streptococcus pneumoniae |
| | 485 + 041.2 | Bronchopneumonia, organism<br>unspecified + pneumococcus | J18.0 + B95.3 | Bronchopneumonia, unspecified organism + Streptococcus pneumoniae |
| Pneumococcal<br>pneumonia | 486 + 041.2 | Pneumonia, organism<br>unspecified + pneumococcus | J18.8 + B95.3<br>J18.9 + B95.3 | Other pneumonia, unspecified organism + Streptococcus pneumoniae<br>Pneumonia, unspecified organism + Streptococcus pneumoniae |
| | 510.x +<br>041.2 | Empyema + pneumococcus | | |
| | 510 + 041.2 | Empyema with fistula +<br>pneumococcus | J86.0 + B95.3 | Pyothorax with fistula + Streptococcus pneumoniae |
| | 510.9 +<br>041.2 | Empyema without mention of<br>fistula + pneumococcus | J86.9 + B95.3 | Pyothorax without fistula + Streptococcus pneumoniae |
| | 480-486<br>487.0 | | Viral, ba | cterial, unspecified pneumonia |
| | 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| Pneumonia<br>with | 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| unspecified<br>causes | 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |
| | 486 | Pneumonia, organism<br>unspecified | J18.8<br>J18.9 | Other pneumonia, unspecified organism Pneumonia, unspecified organism |

Table 4. Diagnosis Codes for Identifying Invasive Pneumococcal Disease, All-Cause Pneumonia, and Pneumococcal Pneumonia

| | | ICD-9-CM | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| IPD | | | | |
| | 790.7 + 041.2<br>771.83 +<br>041.2 | Bacteremia + pneumococcus | R78.81 + B95.3 | Bacteremia + Streptococcus pneumoniae as the cause of diseases classified elsewhere (Streptococcus pneumoniae) |
| Bacteremia | 038.2 | Pneumococcal septicemia | A40.3 | Sepsis due to Streptococcus pneumoniae |
| | 038.9 + 041.2 | Unspecified septicemia +<br>pneumococcus | A41.9 + B95.3 | Sepsis, unspecified organism + Streptococcus pneumoniae |
| | 320.1 | Pneumococcal meningitis | G00.1 | Pneumococcal meningitis |
| Meningitis | 320.9 + 041.2 | Meningitis due to unspecified bacterium + pneumococcus | G00.9 + B95.3<br>G04.2 + B95.3 | Bacterial meningitis, unspecified + Streptococcus pneumoniae<br>Bacterial meningoencephalitis and meningomyelitis, not elsewhere classified +<br>Streptococcus pneumoniae |
| | 322.9 + 041.2 | Meningitis, unspecified +<br>pneumococcus | G03.9 + B95.3 | Meningitis, unspecified + Streptococcus pneumoniae |
| | 421.x + 041.2 | | Endo | ocarditis + pneumococcus |
| | 421 + 041.2 | Acute and subacute bacterial<br>endocarditis + pneumococcus | I33.0 + B95.3 | Acute and subacute infective endocarditis + Streptococcus pneumoniae |
| | 421.1 + 041.2 | Acute and subacute infective<br>endocarditis in diseases<br>classified elsewhere +<br>pneumococcus | I39 + B95.3 | Endocarditis and heart valve disorders in diseases classified elsewhere +<br>Streptococcus pneumoniae |
| Other | 421.9 + 041.2 | Acute endocarditis,<br>unspecified + pneumococcus | I33.9 + B95.3 | Acute and subacute endocarditis, unspecified + Streptococcus pneumoniae |
| | 711.0 + 041.2 | Septic arthritis + pneumococcus | M00.00 + B95.3<br>M00.20 + B95.3<br>M00.80 + B95.3<br>M00.9 + B95.3<br>M00.10 + B95.3 | Staphylococcal arthritis, unspecified joint + Streptococcus pneumoniae Other streptococcal arthritis, unspecified joint + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified joint + Streptococcus pneumoniae Pyogenic arthritis, unspecified + Streptococcus pneumoniae Pneumococcal arthritis, unspecified joint + Streptococcus pneumoniae |

| | | M00.011 + B95.3 | Staphylococcal arthritis, right shoulder + Streptococcus pneumoniae |
|---|---|---|---|
| | | M00.012 + B95.3 | Staphylococcal arthritis, left shoulder + Streptococcus pneumoniae |
| | | M00.019 + B95.3 | Staphylococcal arthritis, unspecified shoulder + Streptococcus pneumoniae |
| | | M00.211 + B95.3 | Other streptococcal arthritis, right shoulder + Streptococcus pneumoniae |
| | | M00.212 + B95.3 | Other streptococcal arthritis, left shoulder + Streptococcus pneumoniae |
| 711.01 + | Pyogenic arthritis, shoulder | M00.219 + B95.3 | Other streptococcal arthritis, unspecified shoulder + Streptococcus pneumoniae |
| 041.2 | region + pneumococcus | M00.811 + B95.3 | Arthritis due to other bacteria, right shoulder + Streptococcus pneumoniae |
| | | M00.812 + B95.3 | Arthritis due to other bacteria, left shoulder + Streptococcus pneumoniae |
| | | M00.819 + B95.3 | Arthritis due to other bacteria, unspecified shoulder + Streptococcus pneumoniae |
| | | M00.119 + B95.3 | Pneumococcal arthritis, unspecified shoulder + Streptococcus pneumoniae |
| | | M00.111 + B95.3 | Pneumococcal arthritis, right shoulder + Streptococcus pneumoniae |
| | | M00.112 + B95.3 | Pneumococcal arthritis, left shoulder + Streptococcus pneumoniae |
| | | M00.021 + B95.3 | Staphylococcal arthritis, right elbow + Streptococcus pneumoniae |
| | | M00.022 + B95.3 | Staphylococcal arthritis, left elbow + Streptococcus pneumoniae |
| | | M00.029 + B95.3 | Staphylococcal arthritis, unspecified elbow + Streptococcus pneumoniae |
| | | M00.221 + B95.3 | Other streptococcal arthritis, right elbow + Streptococcus pneumoniae |
| | | M00.222 + B95.3 | Other streptococcal arthritis, left elbow + Streptococcus pneumoniae |
| 711.02 + | Pyogenic arthritis, upper arm | M00.229 + B95.3 | Other streptococcal arthritis, unspecified elbow + Streptococcus pneumoniae |
| 041.2 | + pneumococcus | M00.821 + B95.3 | Arthritis due to other bacteria, right elbow + Streptococcus pneumoniae |
| | | M00.822 + B95.3 | Arthritis due to other bacteria, left elbow + Streptococcus pneumoniae |
| | | M00.829 + B95.3 | Arthritis due to other bacteria, unspecified elbow + Streptococcus pneumoniae |
| | | M00.129 + B95.3 | Pneumococcal arthritis, unspecified elbow + Streptococcus pneumoniae |
| | | M00.121 + B95.3 | Pneumococcal arthritis, right elbow + Streptococcus pneumoniae |
| | | M00.122 + B95.3 | Pneumococcal arthritis, left elbow + Streptococcus pneumoniae |
| | | M00.031 + B95.3 | Staphylococcal arthritis, right wrist + Streptococcus pneumoniae |
| | | M00.032 + B95.3 | Staphylococcal arthritis, left wrist + Streptococcus pneumoniae |
| | | M00.039 + B95.3 | Staphylococcal arthritis, unspecified wrist + Streptococcus pneumoniae |
| | | M00.231 + B95.3 | Other streptococcal arthritis, right wrist + Streptococcus pneumoniae |
| | | M00.232 + B95.3 | Other streptococcal arthritis, left wrist + Streptococcus pneumoniae |
| 711.03 + | Pyogenic arthritis, forearm + | M00.239 + B95.3 | Other streptococcal arthritis, unspecified wrist + Streptococcus pneumoniae |
| 041.2 | pneumococcus | M00.831 + B95.3 | Arthritis due to other bacteria, right wrist + Streptococcus pneumoniae |
| | | M00.832 + B95.3 | Arthritis due to other bacteria, left wrist + Streptococcus pneumoniae |
| | | M00.839 + B95.3 | Arthritis due to other bacteria, unspecified wrist + Streptococcus pneumoniae |
| | | M00.139 + B95.3 | Pneumococcal arthritis, unspecified wrist + Streptococcus pneumoniae |
| | | M00.131 + B95.3 | Pneumococcal arthritis, right wrist + Streptococcus pneumoniae |
| | | M00.132 + B95.3 | Pneumococcal arthritis, left wrist + Streptococcus pneumoniae |
| | | M00.041 + B95.3 | Staphylococcal arthritis, right hand + Streptococcus pneumoniae |
| | | M00.042 + B95.3 | Staphylococcal arthritis, left hand + Streptococcus pneumoniae |
| 711.04 + | Pyogenic arthritis, hand + | M00.049 + B95.3 | Staphylococcal arthritis, unspecified hand + Streptococcus pneumoniae |
| 041.2 | pneumococcus | M00.241 + B95.3 | Other streptococcal arthritis, right hand + Streptococcus pneumoniae |
| V-1.2 | phemiococcus | M00.242 + B95.3 | Other streptococcal arthritis, left hand + Streptococcus pneumoniae |
| | | M00.249 + B95.3 | Other streptococcal arthritis, unspecified hand + Streptococcus pneumoniae |
| | | M00.841 + B95.3 | Arthritis due to other bacteria, right hand + Streptococcus pneumoniae |
| | | DETAILS CONTENDED | |

| | | M00.842 + B95.3<br>M00.849 + B95.3<br>M00.149 + B95.3<br>M00.141 + B95.3<br>M00.142 + B95.3 | Arthritis due to other bacteria, left hand + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified hand + Streptococcus pneumoniae Pneumococcal arthritis, unspecified hand + Streptococcus pneumoniae Pneumococcal arthritis, right hand + Streptococcus pneumoniae Pneumococcal arthritis, left hand + Streptococcus pneumoniae |
|---|---|---|---|
| 711.05 +<br>041.2 | Pyogenic arthritis, pelvic<br>region and thigh +<br>pneumococcus | M00.051 + B95.3<br>M00.052 + B95.3<br>M00.059 + B95.3<br>M00.251 + B95.3<br>M00.252 + B95.3<br>M00.259 + B95.3<br>M00.851 + B95.3<br>M00.852 + B95.3<br>M00.859 + B95.3<br>M00.159 + B95.3<br>M00.151 + B95.3<br>M00.152 + B95.3 | Staphylococcal arthritis, right hip + Streptococcus pneumoniae Staphylococcal arthritis, left hip + Streptococcus pneumoniae Staphylococcal arthritis, unspecified hip + Streptococcus pneumoniae Other streptococcal arthritis, right hip + Streptococcus pneumoniae Other streptococcal arthritis, left hip + Streptococcus pneumoniae Other streptococcal arthritis, unspecified hip + Streptococcus pneumoniae Arthritis due to other bacteria, right hip + Streptococcus pneumoniae Arthritis due to other bacteria, left hip + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified hip + Streptococcus pneumoniae Pneumococcal arthritis, unspecified hip + Streptococcus pneumoniae Pneumococcal arthritis, inght hip + Streptococcus pneumoniae Pneumococcal arthritis, left hip + Streptococcus pneumoniae |
| 711.06 +<br>041.2 | Pyogenic arthritis, lower leg + pneumococcus | M00.061 + B95.3<br>M00.062 + B95.3<br>M00.069 + B95.3<br>M00.261 + B95.3<br>M00.262 + B95.3<br>M00.269 + B95.3<br>M00.861 + B95.3<br>M00.862 + B95.3<br>M00.869 + B95.3<br>M00.169 + B95.3<br>M00.161 + B95.3<br>M00.162 + B95.3 | Staphylococcal arthritis, right knee + Streptococcus pneumoniae Staphylococcal arthritis, left knee + Streptococcus pneumoniae Staphylococcal arthritis, unspecified knee + Streptococcus pneumoniae Other streptococcal arthritis, right knee + Streptococcus pneumoniae Other streptococcal arthritis, left knee + Streptococcus pneumoniae Other streptococcal arthritis, unspecified knee + Streptococcus pneumoniae Arthritis due to other bacteria, right knee + Streptococcus pneumoniae Arthritis due to other bacteria, left knee + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified knee + Streptococcus pneumoniae Pneumococcal arthritis, unspecified knee + Streptococcus pneumoniae Pneumococcal arthritis, left knee + Streptococcus pneumoniae Pneumococcal arthritis, left knee + Streptococcus pneumoniae |
| 711.07 +<br>041.2 | Pyogenic arthritis, ankle and<br>foot + pneumococcus | M00.071 + B95.3<br>M00.072 + B95.3<br>M00.079 + B95.3<br>M00.271 + B95.3<br>M00.272 + B95.3<br>M00.279 + B95.3<br>M00.871 + B95.3<br>M00.872 + B95.3<br>M00.879 + B95.3<br>M00.179 + B95.3<br>M00.179 + B95.3<br>M00.171 + B95.3 | Staphylococcal arthritis, right ankle and foot + Streptococcus pneumoniae Staphylococcal arthritis, left ankle and foot + Streptococcus pneumoniae Staphylococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, right ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, left ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, right ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, left ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified ankle and foot + Streptococcus pneumoniae Pneumococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae |

| | | | | Pneumococcal arthritis, right ankle and foot + Streptococcus pneumoniae Pneumococcal arthritis, left ankle and foot + Streptococcus pneumoniae |
|---|---|---|---|---|
| | 11.08 +<br>041.2 | Pyogenic arthritis, other<br>specified sites +<br>pneumococcus | M00.08 + B95.3<br>M00.28 + B95.3<br>M00.88 + B95.3<br>M00.9+ B95.3<br>M00.18 + B95.3 | .Staphylococcal arthritis, vertebrae + Streptococcus pneumoniae Other streptococcal arthritis, vertebrae + Streptococcus pneumoniae Arthritis due to other bacteria, vertebrae + Streptococcus pneumoniae Pyogenic arthritis, unspecified + Streptococcus pneumoniae Pneumococcal arthritis, vertebrae + Streptococcus pneumoniae |
| | 11.09 +<br>041.2 | Pyogenic arthritis, multiple<br>sites + pneumococcus | M00.09 + B95.3<br>M00.29 + B95.3<br>M00.89 + B95.3<br>M00.19 + B95.3 | Staphylococcal polyarthritis + Streptococcus pneumoniae Other streptococcal polyarthritis + Streptococcus pneumoniae Polyarthritis due to other bacteria + Streptococcus pneumoniae Pneumococcal polyarthritis + Streptococcus pneumoniae |
| 73 | 30.0x +<br>041.2<br>30.2x +<br>041.2 | | Osteo | omyelitis + pneumococcus |
| | 30.00 +<br>041.2 | Acute osteomyelitis, site unspecified + pneumococcus | M86.00 + B95.3<br>M86.10 + B95.3<br>M86.20 + B95.3 | Acute hematogenous osteomyelitis, unspecified site + Streptococcus pneumoniae Other acute osteomyelitis, unspecified site + Streptococcus pneumoniae Subacute osteomyelitis, unspecified site + Streptococcus pneumoniae |
| | 30.01 +<br>041.2 | Acute osteomyelitis, shoulder region + pneumococcus | M86.011 + B95.3<br>M86.012 + B95.3<br>M86.019 + B95.3<br>M86.111 + B95.3<br>M86.112 + B95.3<br>M86.119 + B95.3<br>M86.211 + B95.3<br>M86.212 + B95.3<br>M86.219 + B95.3 | Acute hematogenous osteomyelitis, right shoulder + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left shoulder + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified shoulder + Streptococcus pneumoniae Other acute osteomyelitis, right shoulder + Streptococcus pneumoniae Other acute osteomyelitis, left shoulder + Streptococcus pneumoniae Other acute osteomyelitis, unspecified shoulder + Streptococcus pneumoniae Subacute osteomyelitis, right shoulder + Streptococcus pneumoniae Subacute osteomyelitis, unspecified shoulder + Streptococcus pneumoniae Subacute osteomyelitis, unspecified shoulder + Streptococcus pneumoniae |
| | 30.02 +<br>041.2 | Acute osteomyelitis, upper arm + pneumococcus | M86.021 + B95.3<br>M86.022 + B95.3<br>M86.029 + B95.3<br>M86.121 + B95.3 | Acute hematogenous osteomyelitis, right humerus + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left humerus + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified humerus + Streptococcus pneumoniae |

| | M96 122 ± D05 2 | Other soute esteeminalitie right humanus + Strantonogue |
|---|---|---|
| | M86.122 + B95.3<br>M86.129 + B95.3<br>M86.221 + B95.3<br>M86.222 + B95.3<br>M86.229 + B95.3 | Other acute osteomyelitis, right humerus + Streptococcus pneumoniae Other acute osteomyelitis, left humerus + Streptococcus pneumoniae Other acute osteomyelitis, unspecified humerus + Streptococcus pneumoniae Subacute osteomyelitis, right humerus + Streptococcus pneumoniae Subacute osteomyelitis, left humerus + Streptococcus pneumoniae Subacute osteomyelitis, unspecified humerus + Streptococcus pneumoniae |
| Acute osteomyelitis, forearm | M86.031 + B95.3<br>M86.032 + B95.3<br>M86.039 + B95.3<br>M86.131 + B95.3<br>M86.132 + B95.3<br>M86.139 + B95.3<br>M86.231 + B95.3<br>M86.232 + B95.3<br>M86.239 + B95.3 | Acute hematogenous osteomyelitis, right radius and ulna + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left radius and ulna + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae Other acute osteomyelitis, right radius and ulna + Streptococcus pneumoniae Other acute osteomyelitis, left radius and ulna + Streptococcus pneumoniae Other acute osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, right radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae |
| Acute osteomyelitis, hand + pneumococcus | M86.041 + B95.3<br>M86.042 + B95.3<br>M86.049 + B95.3<br>M86.141 + B95.3<br>M86.142 + B95.3<br>M86.149 + B95.3<br>M86.241 + B95.3<br>M86.242 + B95.3<br>M86.249 + B95.3 | Acute hematogenous osteomyelitis, right hand + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left hand + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified hand + Streptococcus pneumoniae Other acute osteomyelitis, right hand + Streptococcus pneumoniae Other acute osteomyelitis, left hand + Streptococcus pneumoniae Other acute osteomyelitis, unspecified hand + Streptococcus pneumoniae Subacute osteomyelitis, right hand + Streptococcus pneumoniae Subacute osteomyelitis, left hand + Streptococcus pneumoniae Subacute osteomyelitis, unspecified hand + Streptococcus pneumoniae |
| Acute osteomyelitis, pelvic<br>region and thigh +<br>pneumococcus | M86.051 + B95.3<br>M86.052 + B95.3<br>M86.059 + B95.3<br>M86.151 + B95.3<br>M86.152 + B95.3<br>M86.159 + B95.3<br>M86.251 + B95.3<br>M86.252 + B95.3<br>M86.259 + B95.3 | Acute hematogenous osteomyelitis, right femur + Streptococcus pneumonia Acute hematogenous osteomyelitis, left femur + Streptococcus pneumonia Acute hematogenous osteomyelitis, unspecified femur + Streptococcus pneumonia Other acute osteomyelitis, right femur + Streptococcus pneumonia Other acute osteomyelitis, left femur + Streptococcus pneumonia Other acute osteomyelitis, unspecified femur + Streptococcus pneumonia Subacute osteomyelitis, right femur + Streptococcus pneumoniae Subacute osteomyelitis, left femur + Streptococcus pneumoniae Subacute osteomyelitis, unspecified femur + Streptococcus pneumoniae |
| Acute osteomyelitis, lower leg<br>+ pneumococcus | M86.061 + B95.3<br>M86.062 + B95.3<br>M86.069 + B95.3<br>M86.161 + B95.3 | Acute hematogenous osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae |
| | Acute osteomyelitis, hand + pneumococcus Acute osteomyelitis, pelvic region and thigh + pneumococcus Acute osteomyelitis, lower leg | M86.221 + B95.3 M86.222 + B95.3 M86.229 + B95.3 M86.229 + B95.3 M86.031 + B95.3 M86.032 + B95.3 M86.039 + B95.3 M86.131 + B95.3 M86.132 + B95.3 M86.132 + B95.3 M86.231 + B95.3 M86.232 + B95.3 M86.232 + B95.3 M86.232 + B95.3 M86.241 + B95.3 M86.042 + B95.3 M86.141 + B95.3 M86.141 + B95.3 M86.142 + B95.3 M86.242 + B95.3 M86.242 + B95.3 M86.249 + B95.3 M86.249 + B95.3 M86.251 + B95.3 M86.151 + B95.3 M86.151 + B95.3 M86.152 + B95.3 M86.152 + B95.3 M86.153 + B95.3 M86.154 + B95.3 M86.154 + B95.3 M86.155 + B95.3 M86.155 + B95.3 M86.159 + B95.3 M86.251 + B95.3 M86.252 + B95.3 M86.252 + B95.3 M86.253 + B95.3 M86.254 + B95.3 M86.254 + B95.3 M86.255 + B95.3 M86.256 + B95.3 |

| | | M86.162 + B95.3<br>M86.169 + B95.3<br>M86.261 + B95.3<br>M86.262 + B95.3<br>M86.269 + B95.3 | Other acute osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Other acute osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Other acute osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae |
|---|---|---|---|
| 730.07 +<br>041.2 | Acute osteomyelitis, ankle and foot + pneumococcus | M86.071 + B95.3<br>M86.072 + B95.3<br>M86.079 + B95.3<br>M86.171 + B95.3<br>M86.172 + B95.3<br>M86.179 + B95.3<br>M86.271 + B95.3<br>M86.272 + B95.3<br>M86.279 + B95.3 | Acute hematogenous osteomyelitis, right ankle and foot + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left ankle and foot + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, right ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, left ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, right ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, left ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae |
| 730.08 +<br>041.2 | Acute osteomyelitis, other<br>specified sites +<br>pneumococcus | M86.08 + B95.3<br>M86.18 + B95.3<br>M86.28 + B95.3 | Acute hematogenous osteomyelitis, other sites + Streptococcus pneumoniae Other acute osteomyelitis, other site + Streptococcus pneumoniae Subacute osteomyelitis, other site + Streptococcus pneumoniae |
| 730.09 +<br>041.2 | Acute osteomyelitis, multiple sites<br>+ pneumococcus | M86.09 + B95.3<br>M86.19 + B95.3<br>M86.29 + B95.3 | Acute hematogenous osteomyelitis, multiple sites + Streptococcus pneumoniae Other acute osteomyelitis, multiple sites + Streptococcus pneumoniae Subacute osteomyelitis, multiple sites + Streptococcus pneumoniae |
| 730.2 + 041.2<br>730.21 +<br>041.2<br>730.22 +<br>041.2<br>730.23 +<br>041.2<br>730.24 +<br>041.2<br>730.25 +<br>041.2<br>730.26 +<br>041.2<br>730.27 +<br>041.2<br>730.29 +<br>041.2 | Unspecified osteomyelitis, site unspecified + pneumococcus Unspecified osteomyelitis, shoulder region + pneumococcus Unspecified osteomyelitis, upper arm + pneumococcus Unspecified osteomyelitis, forearm + pneumococcus Unspecified osteomyelitis, hand + pneumococcus Unspecified osteomyelitis, pelvic region and thigh + pneumococcus Unspecified osteomyelitis, lower leg + pneumococcus Unspecified osteomyelitis, ankle and foot + pneumococcus Unspecified osteomyelitis, multiple sites + pneumococcus | M86.9 + B95.3 | Osteomyelitis, unspecified + Streptococcus pneumoniae |

| | 730.28 +<br>041.2 | Unspecified osteomyelitis,<br>other specified sites +<br>pneumococcus | M46.20 + B95.3<br>M46.21 + B95.3<br>M46.22 + B95.3<br>M46.23 + B95.3<br>M46.24 + B95.3<br>M46.25 + B95.3<br>M46.26 + B95.3<br>M46.27 + B95.3<br>M46.28 + B95.3 | Osteomyelitis of vertebra, site unspecified + Streptococcus pneumoniae Osteomyelitis of vertebra, occipito-atlanto-axial region + Streptococcus pneumoniae Osteomyelitis of vertebra, cervical region + Streptococcus pneumoniae Osteomyelitis of vertebra, cervicothoracic region + Streptococcus pneumoniae Osteomyelitis of vertebra, thoracic region + Streptococcus pneumoniae Osteomyelitis of vertebra, thoraciclumbar region + Streptococcus pneumoniae Osteomyelitis of vertebra, lumbar region + Streptococcus pneumoniae Osteomyelitis of vertebra, lumbosacral region + Streptococcus pneumoniae Osteomyelitis of vertebra, sacral and sacrococcygeal region + Streptococcus pneumoniae |
|---|---|---|---|---|
| Pneumonia | | | | |
| | 480-486<br>487.0 | | Viral, ba | cterial, unspecified pneumonia |
| | 480 | Pneumonia due to adenovirus | J12.0 | Adenoviral pneumonia |
| | 480.1 | Pneumonia due to respiratory<br>syncytial virus | J12.1 | Respiratory syncytial virus pneumonia |
| | 480.2 | Pneumonia due to<br>parainfluenza virus | J12.2 | Parainfluenza virus pneumonia |
| | 480.3 | Pneumonia due to SARS-<br>associated coronavirus | J12.81<br>J12.82 | Pneumonia due to SARS-associated coronavirus Pneumonia due to coronavirus disease 2019 |
| | 480.8 | Pneumonia due to other virus<br>not elsewhere classified | J12.3<br>J12.89 | Human metapneumovirus pneumonia<br>Other viral pneumonia |
| | 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| All-Cause | 481 | Pneumococcal pneumonia<br>[Streptococcus pneumoniae<br>pneumonia] | J18.1<br>J13 | Lobar pneumonia, unspecified organism Pneumonia due to Streptococcus pneumoniae |
| | 482 | Pneumonia due to Klebsiella<br>pneumoniae | J15.0 | Pneumonia due to Klebsiella pneumoniae |
| | 482.1 | Pneumonia due to<br>Pseudomonas | J15.1 | Pneumonia due to Pseudomonas |
| | 482.2 | Pneumonia due to Hemophilus<br>influenzae [H. influenzae] | J14 | Pneumonia due to Hemophilus influenzae |
| | 482.3 | Pneumonia due to<br>Streptococcus, unspecified | J15.4 | Pneumonia due to other streptococci |
| | 482.31 | Pneumonia due to<br>Streptococcus, group A | J15.4 | Pneumonia due to other streptococci |
| | 482.32 | Pneumonia due to<br>Streptococcus, group B | J15.3 | Pneumonia due to streptococcus, group B |
| | 482.39 | Pneumonia due to other<br>Streptococcus | J15.4 | Pneumonia due to other streptococci |

| 482.4 | Pneumonia due to<br>Staphylococcus, unspecified | J15.20 | Pneumonia due to staphylococcus, unspecified |
|---|---|---|---|
| 482.41 | Methicillin susceptible<br>pneumonia due to<br>Staphylococcus aureus | J15.211 | Pneumonia due to Methicillin susceptible Staphylococcus aureus |
| 482.42 | Methicillin resistant<br>pneumonia due to<br>Staphylococcus aureus | J15.212 | Pneumonia due to Methicillin resistant Staphylococcus aureus |
| 482.49 | Other Staphylococcus<br>pneumonia | J15.29 | Pneumonia due to other staphylococcus |
| 482.81 | Pneumonia due to anaerobes | J15.8 | Pneumonia due to other specified bacteria |
| 482.82 | Pneumonia due to escherichia<br>coli [E. coli] | J15.5 | Pneumonia due to Escherichia coli |
| 482.83 | Pneumonia due to other gram-<br>negative bacteria | J15.6 | Pneumonia due to other aerobic Gram-negative bacteria |
| 482.84 | Pneumonia due to<br>Legionnaires' disease | A48.1 | Legionnaires' disease |
| 482.89 | Pneumonia due to other<br>specified bacteria | J15.8 | Pneumonia due to other specified bacteria |
| 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| 483 | Pneumonia due to<br>mycoplasma pneumoniae | J15.7 | Pneumonia due to Mycoplasma pneumoniae |
| 483.1 | Pneumonia due to chlamydia | J16.0 | Chlamydial pneumonia |
| 483.8 | Pneumonia due to other<br>specified organism | J16.8 | Pneumonia due to other specified infectious organisms |
| 484.1 | Pneumonia in cytomegalic<br>inclusion disease | B25.0 | Cytomegaloviral pneumonitis |
| 484.3 | Pneumonia in whooping cough | A37.91<br>A37.01<br>A37.11<br>A37.81 | Whooping cough, unspecified species with pneumonia Whooping cough due to Bordetella pertussis with pneumonia Whooping cough due to Bordetella parapertussis with pneumonia Whooping cough due to other Bordetella species with pneumonia |
| 484.5 | Pneumonia in anthrax | A22.1 | Pulmonary anthrax |
| 484.6 | Pneumonia in aspergillosis | B44.0 | Invasive pulmonary aspergillosis |
| 484.7 | Pneumonia in other systemic mycoses | J17 | Pneumonia in diseases classified elsewhere |
| 484.8 | Pneumonia in other infectious<br>diseases classified elsewhere | J17<br>B77.81 | Pneumonia in diseases classified elsewhere<br>Ascariasis pneumonia |
| 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |

| | 486 | Pneumonia, organism<br>unspecified | J18.8<br>J18.9 | Other pneumonia, unspecified organism<br>Pneumonia, unspecified organism |
|---|---|---|---|---|
| | 487 | Influenza with pneumonia | J10.00<br>J10.08<br>J11.00<br>J11.08<br>J12.9 | Influenza due to other identified influenza virus with unspecified type of pneumonia Influenza due to other identified influenza virus with other specified pneumonia Influenza due to unidentified influenza virus with unspecified type of pneumonia Influenza due to unidentified influenza virus with specified pneumonia Viral pneumonia, unspecified |
| | 510.x | | | Empyema |
| | 510 | Empyema with fistula | J86.0 | Pyothorax with fistula |
| | 510.9 | Empyema without mention of fistula | J86.9 | Pyothorax without fistula |
| | | | J85.1 | Abscess of lung with pneumonia |
| | 136.3 | Pneumocystosis | B59 | Pneumocystosis |
| | 481 | Pneumococcal pneumonia | J13 | Pneumonia due to Streptococcus pneumoniae |
| | 482.9 + 041.2 | Bacterial pneumonia,<br>unspecified + pneumococcus | J15.9 + B95.3 | Unspecified bacterial pneumonia + Streptococcus pneumoniae |
| | 485 + 041.2 | Bronchopneumonia, organism<br>unspecified + pneumococcus | J18.0 + B95.3 | Bronchopneumonia, unspecified organism + Streptococcus pneumoniae |
| Pneumococca<br>1 | 486 + 041.2 | Pneumonia, organism<br>unspecified + pneumococcus | J18.8 + B95.3<br>J18.9 + B95.3 | Other pneumonia, unspecified organism + Streptococcus pneumoniae<br>Pneumonia, unspecified organism + Streptococcus pneumoniae |
| | 510.x + 041.2 | Empyema + pneumococcus | | |
| | 510 + 041.2 | Empyema with fistula +<br>pneumococcus | J86.0 + B95.3 | Pyothorax with fistula + Streptococcus pneumoniae |
| | 510.9 + 041.2 | Empyema without mention of<br>fistula + pneumococcus | J86.9 + B95.3 | Pyothorax without fistula + Streptococcus pneumoniae |

# Table 6. National Drug Codes and Procedure Codes for Identifying Immunosuppressive Medications (see excel)

# Table 7. National Drug Codes and Procedure Codes for Identifying Influenza Vaccinations (see excel)

Table 8. National Drug Codes and CPT® Codes for Identifying PPSV23 Vaccination

| Code | Туре | Description |
|-------------|------|--------------|
| 90732 | CPT | Pneumovax 23 |
| 00006473900 | NDC | Pneumovax 23 |
| 00006473901 | NDC | Pneumovax 23 |
| 00006473950 | NDC | Pneumovax 23 |
| 00006474100 | NDC | Pneumovax 23 |
| 00006483701 | NDC | Pneumovax 23 |
| 00006483702 | NDC | Pneumovax 23 |
| 00006483703 | NDC | Pneumovax 23 |
| 00006489400 | NDC | Pneumovax 23 |
| 00006489400 | NDC | Pneumovax 23 |
| 00006494300 | NDC | Pneumovax 23 |
| 00006494301 | NDC | Pneumovax 23 |
| 00247040201 | NDC | Pneumovax 23 |
| 50090145200 | NDC | Pneumovax 23 |
| 50090145209 | NDC | Pneumovax 23 |
| 54569141200 | NDC | Pneumovax 23 |
| 54569653800 | NDC | Pneumovax 23 |
| 54868333901 | NDC | Pneumovax 23 |
| 54868333909 | NDC | Pneumovax 23 |
| 54868432000 | NDC | Pneumovax 23 |
| 54868432009 | NDC | Pneumovax 23 |
| 55045354202 | NDC | Pneumovax 23 |
| 00005230931 | NDC | Pnu-Imune 23 |
| 00005230933 | NDC | Pnu-Imune 23 |
| 54868070700 | NDC | Pnu-Imune 23 |

Table 9. CPT® codes to identify CD4 laboratory tests

| Code | Type | Description |
|-------|------|----------------------|
| 86361 | CPT | Absolute CD4 count |
| 86360 | CPT | Absolute CD4 and CD8 |
| | | counts with ratio |

## Table 10. CPT® codes to identify viral load laboratory tests

| Code | Type | Description |
|---|---|---|
| 87534 | CPT | Infectious agent detection by<br>nucleic acid (DNA or<br>RNA); HIV-1, direct probe<br>technique |
| 87535 | CPT | Infectious agent detection by<br>nucleic acid (DNA or<br>RNA), HIV-1, amplified<br>probe technique |
| 87536 | CPT | Infectious agent detection by<br>nucleic acid (DNA or<br>RNA); HIV-1,<br>quantification |

Table 11. Diagnosis Codes for Identifying All-Cause Pneumonia not due to HIV

| | | ICD-9-CM | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| | 480-486<br>487.0 | | Viral, bacterial, unspecified pneumonia | |
| | 480 | Pneumonia due to adenovirus | J12.0 | Adenoviral pneumonia |
| | 480.1 | Pneumonia due to respiratory<br>syncytial virus | J12.1 | Respiratory syncytial virus pneumonia |
| | 480.2 | Pneumonia due to<br>parainfluenza virus | J12.2 | Parainfluenza virus pneumonia |
| | 480.3 | Pneumonia due to SARS-<br>associated coronavirus | J12.81<br>J12.82 | Pneumonia due to SARS-associated coronavirus Pneumonia due to coronavirus disease 2019 |
| | 480.8 | Pneumonia due to other virus<br>not elsewhere classified | J12.3<br>J12.89 | Human metapneumovirus pneumonia<br>Other viral pneumonia |
| | 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| | 481 | Pneumococcal pneumonia<br>[Streptococcus pneumoniae<br>pneumonia] | J18.1<br>J13 | Lobar pneumonia, unspecified organism<br>Pneumonia due to Streptococcus pneumoniae |
| All-Cause | 482 | Pneumonia due to Klebsiella<br>pneumoniae | J15.0 | Pneumonia due to Klebsiella pneumoniae |
| | 482.1 | Pneumonia due to<br>Pseudomonas | J15.1 | Pneumonia due to Pseudomonas |
| | 482.2 | Pneumonia due to Hemophilus<br>influenzae [H. influenzae] | J14 | Pneumonia due to Hemophilus influenzae |
| | 482.3 | Pneumonia due to<br>Streptococcus, unspecified | J15.4 | Pneumonia due to other streptococci |
| | 482.31 | Pneumonia due to<br>Streptococcus, group A | J15.4 | Pneumonia due to other streptococci |
| | 482.32 | Pneumonia due to<br>Streptococcus, group B | J15.3 | Pneumonia due to streptococcus, group B |
| | 482.39 | Pneumonia due to other<br>Streptococcus | J15.4 | Pneumonia due to other streptococci |
| | 482.4 | Pneumonia due to<br>Staphylococcus, unspecified | J15.20 | Pneumonia due to staphylococcus, unspecified |
| | 482.41 | Methicillin susceptible<br>pneumonia due to<br>Staphylococcus aureus | J15.211 | Pneumonia due to Methicillin susceptible Staphylococcus aureus |

| | 482.42 | Methicillin resistant<br>pneumonia due to<br>Staphylococcus aureus | J15.212 | Pneumonia due to Methicillin resistant Staphylococcus aureus |
|---|---|---|---|---|
| Ī | 482.49 | Other Staphylococcus<br>pneumonia | J15.29 | Pneumonia due to other staphylococcus |
| | 482.81 | Pneumonia due to anaerobes | J15.8 | Pneumonia due to other specified bacteria |
| | 482.82 | Pneumonia due to escherichia<br>coli [E. coli] | J15.5 | Pneumonia due to Escherichia coli |
| [ | 482.83 | Pneumonia due to other gram-<br>negative bacteria | J15.6 | Pneumonia due to other aerobic Gram-negative bacteria |
| | 482.84 | Pneumonia due to<br>Legionnaires' disease | A48.1 | Legionnaires' disease |
| [ | 482.89 | Pneumonia due to other<br>specified bacteria | J15.8 | Pneumonia due to other specified bacteria |
| | 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| | 483.1 | Pneumonia due to chlamydia | J16.0 | Chlamydial pneumonia |
| [ | 483.8 | Pneumonia due to other<br>specified organism | J16.8 | Pneumonia due to other specified infectious organisms |
| | 484.3 | Pneumonia in whooping<br>cough | A37.91<br>A37.01<br>A37.11<br>A37.81 | Whooping cough, unspecified species with pneumonia Whooping cough due to Bordetella pertussis with pneumonia Whooping cough due to Bordetella parapertussis with pneumonia Whooping cough due to other Bordetella species with pneumonia |
| Γ | 484.5 | B | A22.1 | Pulmonary anthrax |
| L | 484.3 | Pneumonia in anthrax | J17 | Pneumonia in diseases classified elsewhere |
| | 484.8 | Pneumonia in other infectious diseases classified elsewhere | J17<br>B77.81 | Pneumonia in diseases classified elsewhere<br>Ascariasis pneumonia |
| Ī | 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |
| | 486 | Pneumonia, organism<br>unspecified | J18.8<br>J18.9 | Other pneumonia, unspecified organism Pneumonia, unspecified organism |
| | 487 | Influenza with pneumonia | J10.00<br>J10.08<br>J11.00<br>J11.08<br>J12.9 | Influenza due to other identified influenza virus with unspecified type of pneumonia Influenza due to other identified influenza virus with other specified pneumonia Influenza due to unidentified influenza virus with unspecified type of pneumonia Influenza due to unidentified influenza virus with specified pneumonia Viral pneumonia, unspecified |

| | 510.x | Empyema | | |
|---|---|---|---|---|
| | 510 | Empyema with fistula | J86.0 | Pyothorax with fistula |
| | 510.9 | Empyema without mention of | J86.9 | Pyothorax without fistula |
| 310 | 510.9 | fistula | J85.1 | Abscess of lung with pneumonia |

Table 12. National Drug Codes and CPT® Codes for Identifying Recombinant Zoster Vaccination

| Code | Туре | Description |
|-------------|------|--------------------------|
| 58160082801 | NDC | Shingrix |
| 58160082803 | NDC | Shingrix |
| 50090514700 | NDC | Shingrix |
| 58160081912 | NDC | Shingrix |
| 58160082311 | NDC | Shingrix |
| 50090337200 | NDC | Shingrix |
| 90750 | CPT | Zoster Vaccine |
| | | Recombinant, Adjuvanted, |
| | | Suspension for |
| | | Intramuscular Injection |

## Table 13. National Drug Codes for Identifying Candidiasis Antifungals (see excel)

## Table 14. Diagnosis Codes for Identifying Opportunistic Infections (see excel)

#### ANNEX 1. LIST OF STAND ALONE DOCUMENTS

If there is no document to be listed, delete the table and write "None".

| Number | Document reference<br>number | Date | Title |
|---|---|---|---|
| 1 | 1 | January 24,<br>2023 | Annex Code Tables |

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not required

## ANNEX 3. ADDITIONAL INFORMATION

Not applicable

## **Document Approval Record**

| Document Name: | B1851217 FINAL | PROTOCOL V3.0 | 06Dec2023 |
|----------------|----------------|---------------|-----------|

Document Title: Assessment of 13-valent pneumococcal conjugate vaccine effectiven

ess among people with HIV in the United States

| s | igned By: | Date(GMT) | Signing Capacity |
|-----|-----------|-------------------|-----------------------------|
| PPD | | 11-Dec-2023 17:4 | 5:08 Business Line Approver |
| | | 11-Dec-2023 18:20 | 6:55 Author Approval |